CLINICAL TRIAL: NCT06116838
Title: Effect of Varying Transcutaneous Spinal Cord Stimulation Parameters and Location on Lower Extremity Motor Responses and Comfort
Brief Title: Transcutaneous Spinal Cord Stimulation in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Executive Director, Technology & Innovation Hub (tiHUB); Director, Max Näder Center for Rehabilitation Technologies & Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: STU00219704
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adults
Keywords: Transcutaneous spinal cord stimulation

STUDY DESIGN:
Intervention Model Description: The purpose of these visits is to determine the optimal waveform and stimulation location. In order to make this determination, we will first determine what stimulation waveform allows us to reach Resting Motor Threshold (RMT) with the lowest intensity but it is the most comfortable when walking at higher intensities. We will use a test-retest design comparing neurophysiologic measures while participants receive various combinations of stimulation waveforms, modulation frequencies, and stimulation locations.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Carrier frequency + Waveform (Experimental): Spinally Evoked Motor Potentials (sEMP) will be obtained while stimulating the spinal cord at a single site with single pulses. sEMP are the electromyograph responses of the peripheral muscles to electrical stimulation of the spinal cord. We will test various waveform combinations of biphasic and monophasic waveforms with modulation frequencies of 0-10 kHz. Participants will also ambulate while receiving continuous stimulation of the various waveform combinations to determine what stimulation intensity is comfortable for each combination. The order we complete this testing will be randomized. All participants will perform testing in a different order.
  Interventions: Device: Spinal motor evoked responses (sMERs); Device: Continuous stimulation tolerance
- Stimulation Location (Experimental): Spinally Evoked Motor Potentials (sEMP) will be obtained while stimulating the spinal cord at various stimulation locations with single pulses. sEMP are the electromyograph responses of the peripheral muscles to electrical stimulation of the spinal cord. Participants will also ambulate while receiving continuous stimulation to various stimulation locations to determine what stimulation intensity is comfortable for each location. The order we complete this testing will be randomized. All participants will perform testing in a different order.
  Interventions: Device: Spinal motor evoked responses (sMERs); Device: Continuous stimulation tolerance

INTERVENTIONS:
Device: Spinal motor evoked responses (sMERs) — Spinally Evoked Motor Responses (sMERs) will be obtained while stimulating with single pulses using various stimulation parameters. sMERs are the electromyograph (EMG) responses of the peripheral muscles to electrical stimulation of the spinal cord. sEMP will be used to test the integrity of the motor pathways of the spinal cord. This will be measuring by assessing the EMG responses in the lower limb muscles.
Device: Continuous stimulation tolerance — Participants may receive up to 45 min of locomotion training (treadmill or overground training) with transcutaneous spinal cord stimulation. The goal will be for the investigators to determine what amount of intensity at each stimulation site the individual finds to be comfortable enough that they would be able to receive without pain or discomfort

SUMMARY:
The goal of this study is to understand how transcutaneous spinal cord stimulation (tSCS) waveform, modulation frequency, and stimulation location impact lower extremity muscle activation and participant comfort in adults without neurologic conditions.

DETAILED DESCRIPTION:
Investigators will use a test-retest design comparing neurophysiologic measures while receiving various combinations of stimulation waveforms, modulation frequencies, and stimulation locations to determine the settings which lead to the highest participant tolerance with the lowest lower extremity resting motor thresholds (RMTs).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Able and willing to give written consent and comply with study procedures

Exclusion Criteria:

* History of stroke or neurologic pathologies (such as multiple sclerosis, Alzheimer's disease, Parkinson's disease, etc.)
* Pregnant or nursing
* Skin allergies or irritation; open wounds
* Utilizing a powered, implanted cardiac device for monitoring or supporting heart function (i.e. pacemaker, defibrillator, or LVAD)
* History of seizures or epilepsy
* Active cancer or cancer in remission less than 5 years
* Metal implants in the back or spine
* Painful musculoskeletal dysfunction due to injury or infection
* Unstable cardiorespiratory or metabolic diseases (e.g. cardiac arrhythmia, uncontrolled hypertension, uncontrolled diabetes, or chronic emphysema)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting motor threshold | All study visits (1-10), over the course of up to 5 weeks
  The RMT is the minimum intensity of stimulation required to evoke a motor response in the lower-limb muscles while the subject is at rest.
Continuous stimulation tolerance | All study visits (1-10), over the course of up to 5 weeks
  Participants may receive up to 45 min of locomotion training (treadmill or overground training) with transcutaneous spinal cord stimulation. Participants will report what level of stimulation intensity they consider comfortable or tolerable (rating of less than 8 out of 10 on the Rating of Perceived Discomfort scale)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayarman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States